CLINICAL TRIAL: NCT02089464
Title: Pivotal Phase III, Prospective, Multicenter, Double Blinded, Randomized, Sham Controlled Trial to Determine the Therapeutic Effects of Navigation Guided 1 Hz rTMS Administered to the Contralesional Hemisphere as Adjuvant to Task Oriented Rehabilitation in Patients With Ischemic or Hemorrhagic Stroke
Brief Title: Niche Trial: Navigated Inhibitory rTMS to Contralesional Hemisphere Trial
Acronym: NICHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nexstim Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NX92325
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NBS-rTMS + task-oriented rehabilitation (Active Comparator): NBS-guided rTMS + task-oriented rehabilitation
  Interventions: Device: NBS-guided rTMS; Procedure: Task oriented rehabilitation
- Sham rTMS + task-oriented rehabilitation (Sham Comparator): Sham rTMS + task-oriented rehabilitation
  Interventions: Device: Sham rTMS; Procedure: Task oriented rehabilitation

INTERVENTIONS:
Device: NBS-guided rTMS
  Other Names: Nexstim
  Arms: NBS-rTMS + task-oriented rehabilitation
Device: Sham rTMS
  Arms: Sham rTMS + task-oriented rehabilitation
Procedure: Task oriented rehabilitation

SUMMARY:
A pivotal, prospective, multi-center, randomized, controlled, double-blinded study combining active Nexstim NBS-guided 1Hz rTMS or sham-rTMS targeting the healthy hemisphere with standardized task oriented rehabilitation will be conducted in patients with post-stroke motor impairment. The therapy will be provided for 6 weeks and primary outcome assessed 6 months later.

ELIGIBILITY:
Inclusion Criteria :

* ≥ 18 years of age
* An ischemic or hemorrhagic stroke suffered 3-12 months prior to the study;
* no other known brain abnormalities by history;
* A one-sided stroke resulting in upper extremity paresis
* A Chedoke-McMaster Stroke Assessment arm stage and hand stage of 3-6 for the affected limb

Exclusion Criteria

* Implanted metallic parts of implanted electronic devices, including pacemakers, defibrillators, or implant medication pump;
* Pregnant or trying to become pregnant; Lack of pregnancy established in females of child-bearing potential by a negative urine pregnancy test at screening.
* Active alcohol abuse, illicit drug use or drug abuse or significant mental illness
* Patients suffering from depression as measured by a score of >10 on the Patient Health Questionnaire (PHQ9). For clarity, patients diagnosed with depression which is controlled with stable anti-depressive medication and in whom PHQ9 is <10 are eligible to participate in the trial.
* History of epilepsy, defined as at least two unprovoked seizures occurring greater than 24 hours apart or diagnosis of an epilepsy syndrome, OR a seizure within the last 12 months.
* Any condition that would prevent the subject from giving voluntary informed consent;
* An implanted brain stimulator;
* Any metal in head with the exception of dental work or any ferromagnetic metal elsewhere in the body;
* Enrolled or plans to enroll in an interventional trial during this study;
* Scalp wounds or infections;
* Claustrophobia precluding MRI;
* A fixed contraction deformity in the affected limb that would prevent normal dexterity if patient were neurologically intact;
* Excessive spasticity as indicated by the Modified Ashworth Spasticity (MAS) Scale >2/4 in either elbow flexors, wrist flexors or finger flexors of the affected limb;i
* previous stroke with residual deficits (TIAs not a reason for exclusion);
* premorbid (retrospective) modified Rankin Scale (mRS) score ≥2 of any aetiology;
* a concurrent progressive neurologic disorder, acute coronary syndrome, severe heart disease (NYHA Classification > 3), or other major medical condition,
* confirmed or suspected lower-limb fracture preventing mobilization,
* patients requiring palliative care
* patients planning to undergo any other occupational therapy during the 6 week active treatment period of the trial (see section 5.2 for study schedule) than what is provided in the study
* A recent injection of botulinium toxin to the affected upper limb in the last 3 months, or the need of an injection of botulinum toxin anytime during the study period and follow up.
* A recent injection of phenol to the affected upper limb in the last 6 months, or the need of an injection of phenol anytime during the study period and follow up.
* Ataxia as measured by a score > 1 on item 7 (limb ataxia) of the NIH stroke scale.
* Severe sensory deficits as measured by a score of 2 on item 8 of the NIH stroke scale.
* Severe aphasia as measured by a score of > 2 on item 9 (best language) of the NIH stroke scale.
* Severe neglect as measured by a score of 2 on item 11 (extinction and inattention) of the NIH stroke scale.
* Patients unable to comprehend or follow verbal commands
* Based on PI's or local physician's assessment patient unable to tolerate the trial procedure due to medical condition
* A Mini mental status exam (MMSE) <25.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Harvey, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (12):
- United States (12):
  - Mayo Clinic, Phoenix, Arizona
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Shepherd Rehabilitation Center, Atlanta, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Indiana University Indianapolis, Indianapolis, Indiana
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Columbia Cornell New York Presbyterian Hospital, New York, New York
  - Burke Medical Research Institute, Weill Cornell Neurology, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - TIRR Memorial Hermann Hospital, Houston, Texas

REFERENCES:
- [Result] Harvey RL, Edwards D, Dunning K, Fregni F, Stein J, Laine J, Rogers LM, Vox F, Durand-Sanchez A, Bockbrader M, Goldstein LB, Francisco GE, Kinney CL, Liu CY; NICHE Trial Investigators *. Randomized Sham-Controlled Trial of Navigated Repetitive Transcranial Magnetic Stimulation for Motor Recovery in Stroke. Stroke. 2018 Sep;49(9):2138-2146. doi: 10.1161/STROKEAHA.117.020607. PMID 30354990

RESULTS

PARTICIPANT FLOW:
Groups:
- NBS-rTMS + Task-oriented Rehabilitation: NBS-guided rTMS + task-oriented rehabilitation
  NBS-guided rTMS
  Task oriented rehabilitation
- Sham rTMS + Task-oriented Rehabilitation: Sham rTMS + task-oriented rehabilitation
  Sham rTMS
  Task oriented rehabilitation
Period: Overall Study
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Started | 132 | 67
Completed | 104 | 51
Not Completed | 28 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation | Total
Number analyzed (Participants) | 132 | 67 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (13.3) | 57.6 (12.7) | 58.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 25 | 69
  Male | 88 | 42 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 18 | 45
  Not Hispanic or Latino | 105 | 49 | 154
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 35 | 12 | 47
  White | 83 | 47 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 132 | 67 | 199
Upper Extremity Fugl-Meyer [Mean (Standard Deviation); unit: units on a scale] — Scale minimum 0, maximum 66. Higher values indicate better motor function.
  units on a scale | 34.0 (12.2) | 35.0 (12.5) | 34.3 (12.3)
Arm Research Action Test [Mean (Standard Deviation); unit: units on a scale] — Scale minimum 0, maximum 57. Greater values indicate better motor function
  units on a scale | 27.3 (16.3) | 30.0 (15.8) | 28.2 (16.1)
Wolf Motor Function Test [Mean (Standard Deviation); unit: seconds of time] — Time in seconds to perform test tasks. Shorter time indicates better motor function.
  seconds of time | 32.1 (48.4) | 29.4 (46.8) | 31.2 (48.1)
Chedoke-McMaster Stroke Assessment Hand [Mean (Standard Deviation); unit: units on a scale] — Scale minimum 1, maximum 7. HIgher score indicates better function.
  units on a scale | 4.0 (0.9) | 4.1 (1.0) | 4.0 (0.9)
Chedoke-McMaster Stroke Assessment Arn [Mean (Standard Deviation); unit: units on a scale] — Scale minimum 1, maximum 7. Higher values indicate better motor function.
  units on a scale | 3.5 (0.8) | 3.6 (0.9) | 3.5 (0.9)
NIH Stroke Scale [Mean (Standard Deviation); unit: units on a scale] — Scale is a measure of neurological functioning, with higher scores reflecting greater deficit (minimum 0,maximum 42)
  units on a scale | 2.7 (1.6) | 2.3 (1.9) | 2.6 (1.8)
Stroke Impact Scale [Mean (Standard Deviation); unit: units on a scale] — Score used to detect the consequences of stroke on physical functioning and activities of daily living. The SIS-16 is a 16 item survey that inquires about daily tasks performed over the previous 2 weeks. Scale minimum 16, maximum 80. Higher values indicate better function.
  units on a scale | 63.3 (16.9) | 65.3 (16.0) | 64.7 (16.8)
Patient Health Questionnaire - 9 (PHQ9) [Mean (Standard Deviation); unit: units on a scale] — The possible presence and severity of depression will be assessed using the Patient Health Questionnaire (PHQ9). PHQ9 is a scale with a minimum value 0 and maximum of 27. Higher values indicate more depressed mood.
  units on a scale | 3.5 (2.9) | 3.7 (3.2) | 3.6 (3.0)
EuroQol ED-5Q scale [Mean (Standard Deviation); unit: units on a scale] — The EuroQoL EQ-5D is a visual analog scale scale from 0 (minimum) to 100 (maximum) assessing quality of life. Higher values indicate better quality of life.
  units on a scale | 68.2 (18.4) | 70.4 (17.9) | 68.8 (18.3)

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity Fugl-Meyer Score
Description: Number of Participants with Improvement in Upper Extremity Fugl-Meyer (UEFM) Score at 6 Months Post-treatment equal or exceeding the Minimal Clinically Important Difference (MCID) of 5 points (MCID).
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
Participants | 88 | 43
Statistical Analysis 1: Comparison: NBS-rTMS + Task-oriented Rehabilitation vs Sham rTMS + Task-oriented Rehabilitation; Test type: Superiority; p = 0.76, Chi-squared

2. Secondary Outcome: Arm-Research Action Test (ARAT)
Description: Scale minimum 0, maximum 57. Greater values indicate better motor function.
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
units on a scale | 5.0 (7.7) | 5.0 (10.9)
Statistical Analysis 1: Comparison: NBS-rTMS + Task-oriented Rehabilitation vs Sham rTMS + Task-oriented Rehabilitation; Test type: Superiority; p = 0.80, t-test, 2 sided

3. Secondary Outcome: Wolf Motor Function Test
Description: Time in seconds to perform test tasks. Shorter time indicates better motor function.
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: seconds of time
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
seconds of time | -9.0 (29.5) | -10.6 (36.5)
Statistical Analysis 1: Comparison: NBS-rTMS + Task-oriented Rehabilitation vs Sham rTMS + Task-oriented Rehabilitation; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: NIH Stroke Scale (NIHSS)
Description: Scale is a measure of neurological functioning, with higher scores reflecting greater deficit (minimum 0,maximum 42)
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
units on a scale | -0.4 (1.3) | -0.7 (1.2)
Statistical Analysis 1: Comparison: NBS-rTMS + Task-oriented Rehabilitation vs Sham rTMS + Task-oriented Rehabilitation; Test type: Superiority; p = 0.14, t-test, 2 sided

5. Secondary Outcome: Chedoke-McMaster Stroke Assessment (CMSA)
Description: Scale minimum 1, maximum 7. Higher values indicate better motor function of hand.
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
units on a scale | 0.5 (1.0) | 0.5 (1.1)
Statistical Analysis 1: Comparison: NBS-rTMS + Task-oriented Rehabilitation vs Sham rTMS + Task-oriented Rehabilitation; Test type: Superiority; p = 0.14, t-test, 2 sided

6. Secondary Outcome: Stroke Impact Scale (SIS)
Description: Score used to detect the consequences of stroke on physical functioning and activities of daily living. The SIS-16 is a 16 item survey that inquires about daily tasks performed over the previous 2 weeks. Scale minimum 16, maximum 80. Higher values indicate better function
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
units on a scale | 6.7 (11.6) | 8.7 (14.5)

7. Secondary Outcome: Patient Health Questionnaire (PHQ9)
Description: The possible presence and severity of depression will be assessed using the Patient Health Questionnaire (PHQ9). PHQ9 is a scale with a minimum value 0 and maximum of 27. Higher values indicate more depressed mood
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
units on a scale | -0.2 (3.3) | 0.0 (4.1)
Statistical Analysis 1: Comparison: NBS-rTMS + Task-oriented Rehabilitation vs Sham rTMS + Task-oriented Rehabilitation; Test type: Superiority; p = 0.95, t-test, 2 sided

8. Secondary Outcome: Quality of Life Assessment: EuroQol EQ-5D Scale
Description: The EuroQoL EQ-5D is a visual analog scale scale from 0 (minimum) to 100 (maximum) assessing quality of life. Higher values indicate better quality of life.
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
units on a scale | 7.7 (15.7) | 6.9 (14.7)
Statistical Analysis 1: Comparison: NBS-rTMS + Task-oriented Rehabilitation vs Sham rTMS + Task-oriented Rehabilitation; Test type: Superiority; p = 0.96, t-test, 2 sided

9. Other Pre Specified Outcome: To Assess Safety of Study Device Use, All Serious Adverse Events Will be Recorded and Compared Between Groups
Description: Serious Adverse Events were recorded and their occurrence was compared between treatment arms
Time Frame: Baseline - 6 months post-treatment
Population: Intent to treat
Measure: Number; unit: number of events
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
Number analyzed (Participants) | 132 | 67
number of events | 16 | 10
Statistical Analysis 1: Comparison: NBS-rTMS + Task-oriented Rehabilitation vs Sham rTMS + Task-oriented Rehabilitation; Test type: Superiority; p = 0.63, Chi-squared

ADVERSE EVENTS:
Arm/Group | NBS-rTMS + Task-oriented Rehabilitation | Sham rTMS + Task-oriented Rehabilitation
All-Cause Mortality (participants affected / at risk) | 1/132 | 0/67
Serious Adverse Events (participants affected / at risk) | 11/132 | 7/67
Other Adverse Events (participants affected / at risk) | 30/132 | 15/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NBS-rTMS + Task-oriented Rehabilitation (N=132) | Sham rTMS + Task-oriented Rehabilitation (N=67)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) — Not study device involvement
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombosis in device (General disorders) | 1 (1) | 0 (0) — Not study device
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NBS-rTMS + Task-oriented Rehabilitation (N=132) | Sham rTMS + Task-oriented Rehabilitation (N=67)
Headache (Nervous system disorders) | 5 (7) | 2 (3)
Paresthesia (Nervous system disorders) | 3 (4) | 1 (2)
Fatigue (General disorders) | 4 (5) | 2 (3)
Spasms in hand (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 1 (1)
Increased lacrimation (Eye disorders) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination olfactory (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No